CLINICAL TRIAL: NCT01798277
Title: Ablation Versus Medical Therapy in Patients With Coronary Artery Disease and Sustained Ventricular Tachycardia Randomized Trial (VeTAMed)
Brief Title: Trial Comparing Ablation With Medical Therapy in Patients With Ventricular Tachycardia
Acronym: VeTAMed
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Low Enrolment
Sponsor: Newmarket Electrophysiology Research Group Inc (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NERG-02
Record Dates: First submitted 2013-02-20; First posted 2013-02-25 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Ventricular Tachycardia; Coronary Artery Disease
Keywords: Keywords provided by Newmarket Electrophysiology Research Group Inc:; Ventricular tachycardia; Ventricular tachyarrhythmia; Ablation; Coronary artery disease; Ischemic heart disease; Amiodarone; Sotalol; Anti-Arrhythmia Agents; Therapeutic Uses; Pharmacologic Actions; Additional relevant MeSH terms:; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes; Catheter Ablation, Radiofrequency
MeSH Terms: conditions — Tachycardia, Ventricular; Coronary Artery Disease; Myocardial Ischemia; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes | interventions — Catheter Ablation; Sotalol; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter Ablation (Active Comparator): Radiofrequency ablation procedure
  Interventions: Procedure: Catheter Ablation
- Medical therapy (Active Comparator): Antiarrhythmic drug therapy will include amiodarone or sotalol. Which antiarrhythmic drug will prescribed per patient depends on the observing physician.
  Interventions: Drug: Medical therapy (sotalol or amiodarone)

INTERVENTIONS:
Procedure: Catheter Ablation — Catheter ablation of ventricular tachycardia will employ three-dimensional mapping Fast Anatomical Mapping or CARTOSOUND technology (Biosense Webster Inc.), and the Thermocool Navistar catheter (Biosense Webster Inc.).
  Other Names: Ablation of:; - Ischemic ventricular tachycardia; - Sustained monomorphic ventricular tachycardia; - Clinical ventricular tachycardia; - Hemodynamically stable/unstable ventricular tachycardia
  Arms: Catheter Ablation
Drug: Medical therapy (sotalol or amiodarone) — Patients will be tiered to one of two possible antiarrhythmic drugs (sotalol or amiodarone).
  Other Names: Sotalol - Betapace, Betapace AF, Sotalex, Sotacor
  Arms: Medical therapy

SUMMARY:
This study aims to compare antiarrhythmic drug therapy with catheter ablation using the SmartTOUCH catheter (Biosense Webster Inc.) as treatment for patients with ventricular tachycardia and coronary artery disease

DETAILED DESCRIPTION:
This is a multicenter, randomized prospective cohort study to compare the impact of catheter ablation with antiarrhythmic drug therapy for treating patients with sustained ventricular tachycardia (VT) and coronary artery disease. Patients that meet all inclusion criteria and no exclusion criteria will be recruited to the study cohort. After baseline measurements are taken, patients will be randomized in a 2:1 fashion to either undergo radiofrequency catheter ablation or receive antiarrhythmic drug therapy (amiodarone or sotalol). The in-clinic appointments include: enrollment, baseline, intervention, and follow-up every three months for one year post-ablation. At each follow-up visit, electrogram (ECG) and Holter monitoring tests will be performed to measure any episodes of ventricular tachyarrhythmia. Furthermore, interrogation of the patient's implantable cardioverter defibrillator (ICD) will be performed at all follow-up visits to detect any episodes of ventricular tachyarrhythmia that required antitachycardia pacing (ATP) or shocks.

ELIGIBILITY:
Inclusion Criteria:

* Sustained monomorphic VT (>30 seconds, or requiring appropriate ICD therapy in patients with ICDs)
* Documented ischemic heart disease with no further options for revascularization
* Ability and willingness to give written informed consent to participate in the trial

Exclusion Criteria:

* VT in the setting of metabolic abnormalities or acute ischemia if coronary lesions suitable for revascularization are identified.
* Acute ischemia with eligibility for revascularization
* Significant peripheral arterial disease preventing transvascular access to the left ventricle.
* Patients with arrhythmogenic right ventricular cardiomyopathy (ARVC), hypertrophic cardiomyopathy, Brugada syndrome, Long QT syndromes, dilated cardiomyopathy
* Prior long term therapy with a Class III or Class IC antiarrhythmic agent (longer than 2 weeks)
* Patient is or may be potentially pregnant
* Patient has a mechanical heart valve
* Myocardial infarction within the past 90 days
* Stroke within the past 90 days
* New York Heart Association (NYHA) functional class IV
* Hemorrhagic manifestations, bleeding diathesis, or impairment of hemostasis
* Lesions at risk of clinically significant bleeding (e.g., extensive cerebral infarction within the last 6 months, active peptic ulcer disease with recent bleeding)
* Prior VT ablation procedure
* Contraindication or allergy to contrast media, routine procedural medications or catheter materials
* Contraindications to an interventional procedure
* Life expectancy is less than 6 months
* Incessant or multiple episodes of VT requiring immediate therapy with medications or ablation
* Untreated hypothyroidism or hyperthyroidism (euthyroid or thyroid hrt is acceptable)
* Current enrolment in another investigational drug or device study
* There are other conditions present that the investigator feels would be problematic or would restrict or limit the participation for the patient for the entire study period
* Absolute contraindication to the use of heparin or warfarin
* Documented intra-arterial thrombus, ventricular thrombus, (less than 6 months after detection of thrombus), tumor or other abnormality that precludes catheter introduction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Ventricular Tachycardia | 1 year
  Number of any appropriate ATPs/shocks and/or presentations of sustained (>30sec) VT on Holter or ECG recording at 3, 6, 9 and 12 months after intervention

SECONDARY OUTCOMES:
Time to First Shock/ATP for VT or to First Presentation of Sustained VT | 1 year
  Change in time to first ATP/shock or presentation of sustained (>30sec) VT on Holter or ECG recording at 3, 6, 9 and 12 months after intervention
Total mortality | 1 year
  Change in mortality status at 3, 6, 9 and 12 months after intervention
Sudden cardiac death | 1 year
  Change in sudden cardiac death status at 3, 6, 9 and 12 months after intervention
Syncope | 1 year
  Change in syncope status at 3, 6, 9 and 12 months after intervention
Number of hospitalizations | 1 year
  Change in number of hospitalizations at 3, 6, 9 and 12 months after intervention
QOL measures | 1 year
  Change in QOL measures at 6 and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yaariv Khaykin, MD, Principal Investigator — Newmarket Electrophysiology Research Group